CLINICAL TRIAL: NCT02670785
Title: A Phase 2, Randomized, Multicenter, Double-blind, Vehicle-controlled Study to Evaluate Safety and Efficacy of Three Doses of Estradiol Vaginal Capsule in Postmenopausal Women With Vulvovaginal Atrophy
Brief Title: A Safety and Efficacy Study of Estradiol Vaginal Capsule in Postmenopausal Women With Vulvovaginal Atrophy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Warner Chilcott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EVC-MD-01
Record Dates: First submitted 2016-01-12; First posted 2016-02-02 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Vulvovaginal Atrophy; Menopause; Dyspareunia
MeSH Terms: conditions — Dyspareunia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Estradiol Vaginal Capsule 0.003 mg (Experimental): Administered intravaginally once daily for 2 weeks and then once weekly for 4 weeks
  Interventions: Drug: Estradiol Vaginal Capsule (EVC)
- Estradiol Vaginal Capsule 0.01 mg (Experimental): Administered intravaginally once daily for 2 weeks and then once weekly for 4 weeks
  Interventions: Drug: Estradiol Vaginal Capsule (EVC)
- Estradiol Vaginal Capsule 0.02 mg (Experimental): Administered intravaginally once daily for 2 weeks and then once weekly for 4 weeks
  Interventions: Drug: Estradiol Vaginal Capsule (EVC)
- Placebo (Placebo Comparator): Administered intravaginally once daily for 2 weeks and then once weekly for 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Estradiol Vaginal Capsule (EVC) — Administered intravaginally once daily for 2 weeks and then once weekly for 4 weeks
  Arms: Estradiol Vaginal Capsule 0.003 mg; Estradiol Vaginal Capsule 0.01 mg; Estradiol Vaginal Capsule 0.02 mg
Drug: Placebo — Administered intravaginally once daily for 2 weeks and then once weekly for 4 weeks
  Arms: Placebo

SUMMARY:
This study will access the safety and efficacy of three doses of estradiol vaginal capsules in postmenopausal women with vulvovaginal atrophy.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of vulvovaginal atrophy due to post menopause
* Age ≥ 40 years or if bilateral oophorectomy ≥ 35 years
* Moderate to severe vaginal dryness
* Normal breast exam; if > 40 years
* Vaginal pH > 5.0
* < 5% superficial cells on vaginal wall cytology smear

Exclusion Criteria:

* Known hypersensitivity to estrogen and/or progestin therapy
* Known or suspected premalignant or malignant disease
* Undiagnosed abnormal genital bleeding
* A history of or treatment for significant cardiovascular disease, congestive heart failure, or stroke
* Active or known protein C, protein S, or antithrombin deficient, or other known thrombophilic disorders or thromboembolic events
* Increased frequency/severity headaches with estrogen therapy
* Smokes ≥ 15 cigarettes/day

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2016-02-15 (Actual); Primary Completion 2016-11-14 (Actual); Study Completion 2016-11-14 (Actual)

PRIMARY OUTCOMES:
Change in the percentage of vaginal superficial cells | Baseline (Week 0) to Final Visit (Week 6)
Change in the percentage of vaginal parabasal cells | Baseline (Week 0) to Final Visit (Week 6)
Change in vaginal pH | Baseline (Week 0) to Final Visit (Week 6)

SECONDARY OUTCOMES:
Change in the investigator assessment of VVA measured by scoring the vaginal health in 5 categories using a 4-point scale | Baseline (Week 0) to Final Visit (Week 6)
  Outcome was measured by using a 4-point severity scale with: None=0, Mild=1, Moderate=2, and Severe=3.
Change in subject's self-assessment of vaginal dryness reported as the most bothersome symptom | Baseline (Week 0) to Final Visit (Week 6)
  Outcome was measured by using a 4-point severity scale with: None=0, Mild=1, Moderate=2, and Severe=3.
Change in subject's self-assessment of dyspareunia reported as the most bothersome symptom | Baseline (Week 0) to Final Visit (Week 6)
  Outcome was measured by using a 4-point severity scale with: None=0, Mild=1, Moderate=2, and Severe=3.
Change in subject's self-assessment of dysuria | Baseline (Week 0) to Final Visit (Week 6)
  Outcome was measured by using a 4-point severity scale with: None=0, Mild=1, Moderate=2, and Severe=3.
Change in subject's self-assessment of vaginal and/or vulvar irritation/itching | Baseline (Week 0) to Final Visit (Week 6)
  Outcome was measured by using a 4-point severity scale with: None=0, Mild=1, Moderate=2, and Severe=3.
Change in subject's self-assessment of vaginal dryness in patients where vaginal dryness was not reported as the most bothersome symptom | Baseline (Week 0) to Final Visit (Week 6)
  Outcome was measured by using a 4-point severity scale with: None=0, Mild=1, Moderate=2, and Severe=3.
Change in subject's self-assessment of dyspareunia in patients where dyspareunia was not reported as the most bothersome symptom | Baseline (Week 0) to Final Visit (Week 6)
  Outcome was measured by using a 4-point severity scale with: None=0, Mild=1, Moderate=2, and Severe=3.
Self-assessment by sexually active participants as to the presence or absence of vaginal bleeding | Baseline (Week 0) to Final Visit (Week 6)
  Total number of participants who were sexually active assessed if vaginal bleeding was present or absent.

CONTACTS AND LOCATIONS:
Overall Officials: Vilma Sniukiene, MD, Study Director — Allergan
Locations (20):
- United States (20):
  - Visions Clinical Research-Tucson, Tucson, Arizona
  - Genesis Center for Clinical Research, San Diego, California
  - Coastal Connecticut Research, LLC, New London, Connecticut
  - Women's Medical Research Group, LLC, Clearwater, Florida
  - Radiant Research, Inc., Pinellas Park, Florida
  - Comprehensive Clinical Trials, LLC, West Palm Beach, Florida
  - Fellows Research Alliance, Inc, Savannah, Georgia
  - Beyer Research, Kalamazoo, Michigan
  - Office of R. Garn Mabey, M.D., Las Vegas, Nevada
  - Carolina Women's Research and Wellness Center, Durham, North Carolina
  - Hawthorne Medical Research, Inc., Winston-Salem, North Carolina
  - Rapid Medical Research, Inc., Cleveland, Ohio
  - Women's Health Research, Columbus, Ohio
  - Clinical Research of Philadelphia, LLC, Philadelphia, Pennsylvania
  - Fellows Research Alliance, Inc, Bluffton, South Carolina
  - Radiant Research, Inc., Dallas, Texas
  - Radiant Research, Inc., San Antonio, Texas
  - Virginia Women's Center, Richmond, Virginia
  - Seattle Women's Health, Research, Gynecology, Seattle, Washington
  - North Spokane Women's Clinic, Spokane, Washington